CLINICAL TRIAL: NCT03215706
Title: A Phase 3, Randomized Study of Nivolumab Plus Ipilimumab in Combination With Chemotherapy vs Chemotherapy Alone as First Line Therapy in Stage IV Non-Small Cell Lung Cancer
Brief Title: A Study of Nivolumab and Ipilimumab Combined With Chemotherapy Compared to Chemotherapy Alone in First Line NSCLC
Acronym: CheckMate 9LA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9LA; 2017-001195-35 (EudraCT Number)
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Nivolumab; Carboplatin; Paclitaxel; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module A (Experimental): Chemotherapy/Biologics combined
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Cisplatin
- Module B (Active Comparator): Chemotherapy Combination
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Biological: Ipilimumab — Specified dose on specified day
  Other Names: Yervoy, BMS734016
  Arms: Module A
Biological: Nivolumab — Specified dose on specified day
  Other Names: Opdivo, BMS936558
  Arms: Module A
Drug: Carboplatin — Specified dose on specified day
Drug: Paclitaxel — Specified dose on specified day
  Other Names: Taxol
Drug: Pemetrexed — Specified dose on specified day
  Other Names: Alimta
Drug: Cisplatin — Specified dose on specified day
  Other Names: Platinol

SUMMARY:
The purpose of this study is to determine whether Nivolumab, Ipilimumab combined with chemotherapy is more effective than chemotherapy by itself when treating stage IV NSCLC as the first treatment given for the disease

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants with histologically confirmed Stage IV or recurrent NSCLC squamous or non-squamous histology, with no prior systemic anticancer therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Measurable disease by CT or MRI per response evaluation criteria in solid tumors version 1.1 (RECIST 1.1) criteria
* Participants must have PD-L1 IHC testing with results performed by a central laboratory during the screening period

Exclusion Criteria:

* Participants with known epidermal growth factor receptor (EGFR) mutations which are sensitive to available targeted inhibitor therapy (including, but not limited to, deletions in exon 19 and exon 21 [L858R] substitution mutations) are excluded
* Participants with known anaplastic lymphoma kinase (ALK) translocations which are sensitive to available targeted inhibitor therapy are excluded
* Participants with untreated CNS metastases are excluded. Participants are eligible if CNS metastases are adequately treated and participants are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to first treatment

Other protocol inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (116):
- United States (16):
  - Memorial Health Systems, Colorado Springs, Colorado
  - Local Institution - 0044, Plainville, Connecticut
  - Local Institution - 0045, Jacksonville, Florida
  - Local Institution - 0029, Marietta, Georgia
  - Local Institution - 0091, Wichita, Kansas
  - Local Institution - 0004, Lexington, Kentucky
  - Local Institution - 0105, Detroit, Michigan
  - Local Institution - 0058, Johnson City, New York
  - Local Institution - 0098, Mineola, New York
  - Local Institution - 0095, Columbus, Ohio
  - Local Institution - 0006, Lancaster, Pennsylvania
  - Local Institution - 0047, Pittsburgh, Pennsylvania
  - Local Institution - 0093, Pittsburgh, Pennsylvania
  - Local Institution - 0094, Charleston, South Carolina
  - Southwest Regional Cancer Clinic, St. George, Utah
  - Local Institution - 0099, Madison, Wisconsin
- Argentina (5):
  - Local Institution - 0014, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0028, Río Cuarto, Córdoba Province
  - Local Institution - 0026, Viedma, Río Negro Province
  - Local Institution - 0027, Rosario, Santa Fe Province
  - Local Institution - 0030, Córdoba
- Australia (5):
  - Local Institution - 0086, Gosford, New South Wales
  - Local Institution - 0040, Bedford Park, South Australia
  - Local Institution - 0089, Box Hill, Victoria
  - Local Institution - 0036, Heidelberg, Victoria
  - Local Institution - 0078, Murdoch, Western Australia
- Belgium (3):
  - Local Institution - 0002, Gilly
  - Local Institution - 0033, Leuven
  - Local Institution - 0001, Roeselare
- Brazil (8):
  - Local Institution - 0068, Natal, Rio Grande do Norte
  - Local Institution - 0063, Ijuí, Rio Grande do Sul
  - Local Institution - 0067, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0069, Blumenau, Santa Catarina
  - Local Institution - 0064, Barretos, São Paulo
  - Local Institution - 0065, São José do Rio Preto, São Paulo
  - Local Institution - 0066, Rio de Janeiro
  - Local Institution - 0070, São Paulo
- Canada (4):
  - Local Institution - 0090, Montreal, Quebec
  - Local Institution - 0083, Montreal, Quebec
  - Local Institution - 0082, Montreal, Quebec
  - Local Institution - 0080, Rimouski, Quebec
- Chile (3):
  - Local Institution - 0079, Viña del Mar, Región de Valparaíso
  - Local Institution - 0059, Santiago, Santiago Metropolitan
  - Local Institution - 0084, Santiago, Santiago Metropolitan
- China (11):
  - Local Institution - 0139, Beijing, BEI
  - Local Institution - 0146, Haikou, Hainan
  - Local Institution - 0148, Zhengzhou, Henan
  - Local Institution - 0120, Zhengzhou, Henan
  - Local Institution - 0144, Changsha, Hunan
  - Local Institution - 0106, Changchun, Jilin
  - Local Institution - 0108, Xi'an, Shan3xi
  - Local Institution - 0110, Hangzhou, Zhejiang
  - Local Institution - 0111, Zhejiang, Zhejiang
  - Local Institution - 0113, Beijing
  - Local Institution - 0112, Shanghai
- France (8):
  - Local Institution - 0010, Bron, Auvergne-Rhône-Alpes
  - Local Institution - 0009, Lyon Cedex08, Auvergne-Rhône-Alpes
  - Local Institution - 0013, Caen
  - Local Institution - 0071, Lille
  - Local Institution - 0012, Montpellier
  - Local Institution - 0035, Nantes
  - Local Institution - 0011, Paris
  - Local Institution - 0097, Saint-Brieuc
- Germany (8):
  - Local Institution - 0073, Berlin
  - Local Institution - 0016, Gauting
  - Local Institution - 0072, Großhansdorf
  - Local Institution - 0019, Hemer
  - Local Institution - 0017, Immenhausen
  - Local Institution - 0074, Magdeburg
  - Local Institution - 0015, München
  - Local Institution - 0018, Stuttgart
- Ireland (2):
  - Local Institution - 0021, Dublin
  - Local Institution - 0020, Limerick
- Italy (3):
  - Local Institution - 0042, Lucca
  - Local Institution - 0041, Milan
  - Local Institution - 0043, Napoli
- Japan (21):
  - Local Institution - 0101, Fukushima, Fukushima
  - Local Institution - 0118, Maebashi, Gunma
  - Local Institution - 0128, Ota-shi, Gunma
  - Local Institution - 0138, Hiroshima, Hiroshima
  - Local Institution - 0137, Hiroshima, Hiroshima
  - Local Institution - 0127, Sapporo, Hokkaido
  - Local Institution - 0131, Akashi-shi, Hyōgo
  - Local Institution - 0119, Himeji-shi, Hyōgo
  - Local Institution - 0104, Kobe, Hyōgo
  - Local Institution - 0115, Kanazawa, Ishikawa-ken
  - Local Institution - 0100, Shiwa-gun, Iwate
  - Local Institution - 0129, Yokohama, Kanagawa
  - Local Institution - 0114, Yokohama, Kanagawa
  - Local Institution - 0134, Yokohama, Kanagawa
  - Local Institution - 0116, Niigata, Niigata
  - Local Institution - 0136, Okayama, Okayama-ken
  - Local Institution - 0135, Habikino-shi, Osaka
  - Local Institution - 0103, Ōsaka-sayama, Osaka
  - Local Institution - 0102, Kitaadachi-gun, Saitama
  - Local Institution - 0132, Ube-shi, Yamaguchi
  - Local Institution - 0130, Osaka
- Mexico (3):
  - Local Institution - 0077, La Paz, BAJA Californa SUR
  - Local Institution - 0061, Guadalajara, Jalisco
  - Local Institution - 0075, Veracruz, Veracruz
- Poland (3):
  - Local Institution - 0087, Bydgoszcz
  - Local Institution - 0022, Bytom
  - Local Institution - 0085, Gdansk
- Romania (3):
  - Local Institution - 0034, Bucharest
  - Local Institution - 0031, Cluj-Napoca
  - Local Institution - 0032, Craiova
- Russia (2):
  - Local Institution - 0024, Moscow
  - Local Institution - 0025, Saint Petersburg
- Spain (5):
  - Local Institution - 0054, A Coruña
  - Local Institution - 0053, Barcelona
  - Local Institution - 0052, Madrid
  - Local Institution - 0055, Málaga
  - Local Institution - 0056, Valencia
- United Kingdom (3):
  - Local Institution - 0050, Guildford
  - Local Institution - 0049, London
  - Local Institution - 0048, Tauton

REFERENCES:
- [Derived] Peters S, Paz-Ares LG, Reck M, Carbone DP, Brahmer JR, Borghaei H, Lu S, O'Byrne KJ, John T, Ciuleanu TE, Schenker M, Bernabe Caro R, Nishio M, Cobo M, Lee JS, Zurawski B, Pluzanski A, Aoyama T, Tschaika M, Devas V, Grootendorst DJ, Ramalingam SS. Long-Term Survival Outcomes With First-Line Nivolumab Plus Ipilimumab-Based Treatment in Patients With Metastatic NSCLC and Tumor Programmed Death-Ligand 1 Lower Than 1%: A Pooled Analysis. J Thorac Oncol. 2025 Jan;20(1):94-108. doi: 10.1016/j.jtho.2024.09.1439. Epub 2024 Oct 4. PMID 39369790
- [Derived] Reck M, Ciuleanu TE, Schenker M, Bordenave S, Cobo M, Juan-Vidal O, Reinmuth N, Richardet E, Felip E, Menezes J, Cheng Y, Mizutani H, Zurawski B, Alexandru A, Carbone DP, Lu S, John T, Aoyama T, Grootendorst DJ, Hu N, Eccles LJ, Paz-Ares LG. Five-year outcomes with first-line nivolumab plus ipilimumab with 2 cycles of chemotherapy versus 4 cycles of chemotherapy alone in patients with metastatic non-small cell lung cancer in the randomized CheckMate 9LA trial. Eur J Cancer. 2024 Nov;211:114296. doi: 10.1016/j.ejca.2024.114296. Epub 2024 Aug 25. PMID 39270380
- [Derived] Paz-Ares L, Ciuleanu TE, Cobo M, Schenker M, Zurawski B, Menezes J, Richardet E, Bennouna J, Felip E, Juan-Vidal O, Alexandru A, Sakai H, Lingua A, Salman P, Souquet PJ, De Marchi P, Martin C, Perol M, Scherpereel A, Lu S, John T, Carbone DP, Meadows-Shropshire S, Agrawal S, Oukessou A, Yan J, Reck M. First-line nivolumab plus ipilimumab combined with two cycles of chemotherapy in patients with non-small-cell lung cancer (CheckMate 9LA): an international, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Feb;22(2):198-211. doi: 10.1016/S1470-2045(20)30641-0. Epub 2021 Jan 18. PMID 33476593
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 707 Randomized and treated
Groups:
- Treatment A: Nivolumab + Ipilimumab + Chemotherapy
- Treatment B: Chemotherapy only
Period: Randomization
Arm/Group | Treatment A | Treatment B
Started (= Participants Randomized) | 361 | 358
Completed (= Participants treated) | 358 | 349
Not Completed | 3 | 9
Not completed — Adverse Event unrelated to study drug | 1 | 0
Not completed — participant withdrew consent | 1 | 3
Not completed — no longer meets study criteria | 1 | 4
Not completed — other reasons | 0 | 2
Period: Treatment Period
Arm/Group | Treatment A | Treatment B
Started (= Participants treated) | 358 | 349
Completed (= completing treatment) | 49 | 100
Not Completed | 309 | 249
Not completed — Disease Progression | 184 | 174
Not completed — Study Drug Toxicity | 70 | 24
Not completed — Death | 7 | 1
Not completed — Adverse event unrelated to study drug | 31 | 27
Not completed — Request to D/C treatment | 2 | 10
Not completed — Participant withdrew consent | 4 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative reason by sponsor | 0 | 2
Not completed — other reasons | 10 | 5
Not completed — Not reported | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Total
Number analyzed (Participants) | 361 | 358 | 719
Age, Continuous [Median (Standard Deviation); unit: Years] | 65.0 (8.3) | 65.0 (10.3) | 65.0 (9.4)
Age, Customized [Number; unit: Count of Participants]
  ˂65 years old | 176 | 178 | 49.2
  ≥65 and ˂75 years old | 148 | 147 | 41.0
  ≥75 years old | 37 | 33 | 9.7
  ≥85 years old | 0 | 2 | 0.3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 106 | 215
  Male | 252 | 252 | 504
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 31 | 60
  Not Hispanic or Latino | 154 | 158 | 312
  Unknown or Not Reported | 178 | 169 | 347
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 322 | 316 | 638
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death from any cause. OS was censored on the last date a subject was known to be alive. Survival follow-up was to be conducted every 3 months after participants's off-treatment date.
Time Frame: From date of randomization to date of death (assessed up to October 2019, approximately 23 months)
Population: All Randomized Participants, Global Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 361 | 358
Months | 14.13 [13.24 to 16.16] | 10.74 [9.46 to 12.45]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority — Treatment A over Treatment B; p = 0.0006, Log-rank test stratified; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.56 to 0.86]

2. Secondary Outcome: Progression Free Survival (PFS) by BICR
Description: PFS (primary definition) was defined as the time from the randomization date to the date of the first documented tumor progression based on BICR assessment (per RECIST 1.1), or death from any cause, whichever occurred first. Participants who died without a reported prior progression were considered to have progressed on the date of their death. Participants who had not progressed or died were censored on the date of their last evaluable tumor assessment. Participants who did not have any on-study tumor assessments and did not die were censored on the randomization date. Participants who started any palliative local therapy or subsequent anticancer therapy without a prior reported progression were censored at the last evaluable tumor assessment prior to initiation of the palliative local therapy or subsequent anti-cancer therapy, whichever procedure occurred first.
Time Frame: From date of randomization until date of documented tumor progression or death due to any cause, whichever occurs first (assessed up to October 2024, approximately 72 months)
Population: All Randomized Participants, Global Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 361 | 358
Months | 6.74 [5.55 to 8.05] | 5.26 [4.37 to 5.59]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority — Treatment A over Treatment B; Log-rank test stratified; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.59 to 0.82]

3. Secondary Outcome: Objective Response Rate (ORR) by BICR
Description: ORR was defined as the number of randomized participants with a best overall response (BOR) of confirmed CR or PR based on BICR assessments (using RECIST v1.1 criteria), divided by the number of all randomized participants. BOR was recorded between the date of randomization and the date of objectively documented progression per RECIST 1.1 or the date of initiation of palliative local therapy or the date of initiation of subsequent anti-cancer therapy, whichever occurred first. For participants without documented progression or palliative local therapy or subsequent anti-cancer therapy, all available response designations contributed to the BOR determination. For participants who continued treatment beyond progression, the BOR was determined based on response designations recorded up to the time of the initial RECIST 1.1 defined progression.
Time Frame: as for outcome 2
Population: All Randomized Participants, Global Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 361 | 358
Percentage of Participants | 38.0 [32.9 to 43.2] | 25.1 [20.7 to 30.0]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority — Treatment A over Treatment B; Mantel Haenszel; Odds Ratio (OR) = 12.7, 95% CI 2-sided [6.0 to 19.4]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time between the date of first confirmed documented response (CR or PR) to the date of the first documented BICR-assessed tumor progression (per RECIST 1.1), or death from any cause, whichever occurred first. Participants who started subsequent therapy (including palliative local therapy) without a prior reported progression were censored at the last evaluable tumor assessments prior to initiation of the subsequent anticancer therapy (including palliative local therapy). Participants who died without a reported prior progression were considered to have progressed on the date of their death. For subjects who neither progressed nor died, DoR was censored on the date of their last evaluable tumor assessment. DoR was evaluated for responders (confirmed CR or PR) only.
Time Frame: as for outcome 2
Population: All confirmed Responders, Global Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 137 | 90
Months | 13.01 [8.71 to 20.21] | 5.59 [4.37 to 7.10]

5. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time from randomization to the date of the first confirmed documented response (CR or PR), as assessed by the BICR. TTR was evaluated for responders (confirmed CR or PR) only.
Time Frame: as for outcome 2
Population: All Confirmed Responders, Global Population
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 137 | 90
Months | 2.53 [1.1 to 52.1] | 1.58 [1.2 to 22.2]

6. Secondary Outcome: Objective Response Rate (ORR) by BICR by PD-LI Tumor Cell Expression
Description: ORR was defined as the proportion of randomized participants with a best overall response (BOR) of confirmed complete or partial response per BICR using RECIST v1.1. BOR was assessed from randomization until documented progression, start of palliative local or subsequent anti-cancer therapy-whichever came first. If none occurred, all response data contributed to BOR. For those treated beyond progression, BOR was based on responses before initial RECIST-defined progression. PD-L1 expression was measured via Dako PD-L1 IHC 28-8 pharmDx test as the percentage of tumor cells with membrane staining among ≥100 evaluable cells. Expression was categorized as ≥1%, <1%, not quantifiable, ≥50%, or 1-49%.
Time Frame: as for outcome 2
Population: All Randomized Participants, Global Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 361 | 358
Percentage of Participants
  BASELINE PD-L1 EXPRESSION ≥1%: number analyzed (Participants) | 204 | 204
  BASELINE PD-L1 EXPRESSION ≥1% | 42.6 [35.8 to 49.7] | 27.5 [21.5 to 34.1]
  BASELINE PD-L1 EXPRESSION < 1%: number analyzed (Participants) | 135 | 129
  BASELINE PD-L1 EXPRESSION < 1% | 31.1 [23.4 to 39.6] | 20.2 [13.6 to 28.1]
  Non-Quantifiable PD-L1 Expression: number analyzed (Participants) | 22 | 25
  Non-Quantifiable PD-L1 Expression | 36.4 [17.2 to 59.3] | 32.0 [14.9 to 53.5]
  BASELINE PD-L1 EXPRESSION 1 - 49%: number analyzed (Participants) | 128 | 106
  BASELINE PD-L1 EXPRESSION 1 - 49% | 38.3 [29.8 to 47.3] | 23.6 [15.9 to 32.8]
  BASELINE PD-L1 EXPRESSION >= 50%: number analyzed (Participants) | 76 | 98
  BASELINE PD-L1 EXPRESSION >= 50% | 50.0 [38.3 to 61.7] | 31.6 [22.6 to 41.8]

7. Secondary Outcome: PFS by BICR by PD-L1 Tumor Cell Expression
Description: as for outcome 2
Time Frame: as for outcome 2
Population: All Randomized Participants, Global Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 361 | 358
Months
  < 1% PD-L1 Expression: number analyzed (Participants) | 135 | 129
  < 1% PD-L1 Expression | 5.78 [4.40 to 7.66] | 4.96 [4.21 to 5.78]
  >= 1% PD-L1 Expression: number analyzed (Participants) | 204 | 204
  >= 1% PD-L1 Expression | 6.87 [5.55 to 8.94] | 4.70 [4.24 to 5.55]
  with 1-49% PD-L1 Expression: number analyzed (Participants) | 128 | 106
  with 1-49% PD-L1 Expression | 6.74 [4.50 to 8.51] | 5.29 [4.24 to 5.68]
  with >= 50% PD-L1 Expression: number analyzed (Participants) | 76 | 98
  with >= 50% PD-L1 Expression | 8.28 [4.44 to 12.48] | 4.53 [4.14 to 5.65]
  Non-Quantifiable PD-L1 Expression: number analyzed (Participants) | 22 | 25
  Non-Quantifiable PD-L1 Expression | 6.95 [3.61 to 15.08] | 6.77 [2.83 to 13.83]

8. Secondary Outcome: OS by PD-L1 Tumor Cell Expression
Description: as for outcome 1
Time Frame: From date of randomization to date of death (assessed up to October 2024, approximately 72 months)
Population: All Randomized Participants, Global Population with PD-L1 measurements
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 360 | 358
Months
  < 1% PD-L1 Expression: number analyzed (Participants) | 135 | 129
  < 1% PD-L1 Expression | 17.74 [13.67 to 20.27] | 9.79 [7.69 to 13.54]
  >= 1% PD-L1 Expression: number analyzed (Participants) | 204 | 204
  >= 1% PD-L1 Expression | 15.80 [13.77 to 22.18] | 10.89 [9.49 to 13.17]
  with 1-49% PD-L1 Expression: number analyzed (Participants) | 128 | 106
  with 1-49% PD-L1 Expression | 15.20 [12.62 to 21.22] | 10.37 [8.67 to 12.35]
  with >= 50% PD-L1 Expression: number analyzed (Participants) | 76 | 98
  with >= 50% PD-L1 Expression | 18.91 [13.11 to 29.11] | 12.93 [9.36 to 17.58]
  Non-Quantifiable PD-L1 Expression: number analyzed (Participants) | 21 | 25
  Non-Quantifiable PD-L1 Expression | 10.84 [7.16 to 15.57] | 17.05 [8.64 to NA] — Upper Limit Not Reached

9. Post Hoc Outcome: Overall Survival (OS)
Description: as for outcome 1
Time Frame: From date of randomization to date of death (assessed up to October 2024, approximately 72 months)
Population: All Randomized Participants, Global Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 361 | 358
Months | 15.80 [13.93 to 19.71] | 10.96 [9.49 to 12.71]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority — Treatment A over Treatment B; Stratified Cox proportional hazard model; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.63 to 0.87]

10. Secondary Outcome: PFS by BICR by Tumor Mutational Burden
Description: as for outcome 2
Time Frame: as for outcome 2
Population: All Randomized Participants, Global Population with tumor mutational burden measurements
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 355 | 356
Months
  ≥ 10 Mutations/MB: number analyzed (Participants) | 101 | 82
  ≥ 10 Mutations/MB | 8.94 [5.55 to 13.01] | 4.70 [4.14 to 5.62]
  < 10 Mutations/MB: number analyzed (Participants) | 136 | 137
  < 10 Mutations/MB | 5.62 [4.17 to 7.20] | 5.16 [4.21 to 5.62]
  Overall: number analyzed (Participants) | 237 | 219
  Overall | 6.37 [5.36 to 8.21] | 4.96 [4.27 to 5.55]
  Not Evaluable: number analyzed (Participants) | 118 | 137
  Not Evaluable | 6.74 [4.24 to 9.69] | 5.45 [4.17 to 5.82]

11. Secondary Outcome: ORR by BICR by Tumor Mutational Burden
Description: as for outcome 3
Time Frame: as for outcome 2
Population: All Randomized Participants, Global Population with tumor mutational burden measurements
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 355 | 356
Percentage of Participants
  ≥ 10 Mutations/MB: number analyzed (Participants) | 101 | 82
  ≥ 10 Mutations/MB | 45.5 [35.6 to 55.8] | 29.3 [19.7 to 40.4]
  < 10 Mutations/MB: number analyzed (Participants) | 136 | 137
  < 10 Mutations/MB | 31.6 [23.9 to 40.1] | 27.0 [19.8 to 35.3]
  Overall: number analyzed (Participants) | 237 | 219
  Overall | 37.6 [31.4 to 44.1] | 27.9 [22.0 to 34.3]
  Not Evaluable: number analyzed (Participants) | 118 | 137
  Not Evaluable | 36.4 [27.8 to 45.8] | 21.2 [14.7 to 29.0]

12. Secondary Outcome: OS by Tumor Mutational Burden
Description: as for outcome 1
Time Frame: From date of randomization to date of death (assessed up to October 2024, approximately 72 months)
Population: All Randomized Participants, Global Population with tumor mutational burden measurements
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 355 | 356
Months
  ≥ 10 Mutations/MB: number analyzed (Participants) | 101 | 82
  ≥ 10 Mutations/MB | 15.05 [12.45 to 20.76] | 10.76 [7.85 to 15.41]
  < 10 Mutations/MB: number analyzed (Participants) | 136 | 137
  < 10 Mutations/MB | 16.51 [11.99 to 19.98] | 12.55 [10.38 to 14.92]
  Overall: number analyzed (Participants) | 237 | 219
  Overall | 15.57 [13.34 to 19.38] | 12.06 [10.35 to 14.06]
  Not Evaluable: number analyzed (Participants) | 118 | 137
  Not Evaluable | 17.10 [13.47 to 25.49] | 9.46 [8.15 to 11.79]

ADVERSE EVENTS:
Time Frame: 30 days after last dose, assessed up to October 2024, approximately 72 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Treatment A | Treatment B
All-Cause Mortality (participants affected / at risk) | 304/361 | 318/358
Serious Adverse Events (participants affected / at risk) | 259/358 | 197/349
Other Adverse Events (participants affected / at risk) | 343/358 | 329/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=358) | Treatment B (N=349)
Anaemia (Blood and lymphatic system disorders) | 11 | 18
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 9
Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 7
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 3
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 2 | 1
Cor pulmonale chronic (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericardial effusion malignant (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 7 | 0
Hypophysitis (Endocrine disorders) | 4 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 5 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 3
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 4
Pancreatitis (Gastrointestinal disorders) | 6 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 6
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 2 | 1
Fatigue (General disorders) | 4 | 1
General physical health deterioration (General disorders) | 5 | 5
Illness (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 2
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Mucosal inflammation (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 4 | 1
Pain (General disorders) | 4 | 3
Polyserositis (General disorders) | 1 | 0
Pyrexia (General disorders) | 6 | 1
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 3 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 5 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 0
Hepatotoxicity (Hepatobiliary disorders) | 3 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Contrast media reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Abscess jaw (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 7 | 0
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 3
Clostridial sepsis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Coronavirus pneumonia (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 2 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infective spondylitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 1 | 2
Mastoiditis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 2
Pleural infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 28 | 23
Pneumonia aspiration (Infections and infestations) | 2 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 3 | 5
Sepsis (Infections and infestations) | 3 | 5
Septic shock (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Vascular device infection (Infections and infestations) | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 2 | 0
General physical condition abnormal (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2
Troponin increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 7 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 61 | 78
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Agraphia (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalitis autoimmune (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Immune-mediated encephalitis (Nervous system disorders) | 1 | 0
Medullary compression syndrome (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Quadriplegia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 1
VIth nerve disorder (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Mental status changes (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 8 | 6
Haematuria (Renal and urinary disorders) | 0 | 1
Immune-mediated nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 1
Urinary retention (Renal and urinary disorders) | 1 | 2
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery compression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 2 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=358) | Treatment B (N=349)
Anaemia (Blood and lymphatic system disorders) | 122 | 161
Neutropenia (Blood and lymphatic system disorders) | 39 | 60
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 38
Hyperthyroidism (Endocrine disorders) | 32 | 2
Hypothyroidism (Endocrine disorders) | 61 | 12
Abdominal pain (Gastrointestinal disorders) | 28 | 22
Abdominal pain upper (Gastrointestinal disorders) | 19 | 17
Constipation (Gastrointestinal disorders) | 85 | 83
Diarrhoea (Gastrointestinal disorders) | 111 | 68
Nausea (Gastrointestinal disorders) | 120 | 146
Vomiting (Gastrointestinal disorders) | 71 | 61
Asthenia (General disorders) | 112 | 96
Chest pain (General disorders) | 21 | 8
Fatigue (General disorders) | 81 | 62
Mucosal inflammation (General disorders) | 20 | 10
Oedema peripheral (General disorders) | 28 | 37
Pyrexia (General disorders) | 52 | 39
Bronchitis (Infections and infestations) | 21 | 9
Pneumonia (Infections and infestations) | 24 | 14
Upper respiratory tract infection (Infections and infestations) | 18 | 8
Urinary tract infection (Infections and infestations) | 19 | 11
Alanine aminotransferase increased (Investigations) | 31 | 21
Amylase increased (Investigations) | 38 | 17
Aspartate aminotransferase increased (Investigations) | 30 | 14
Blood alkaline phosphatase increased (Investigations) | 24 | 23
Blood creatinine increased (Investigations) | 26 | 25
Lipase increased (Investigations) | 39 | 9
Neutrophil count decreased (Investigations) | 20 | 12
Platelet count decreased (Investigations) | 14 | 18
Weight decreased (Investigations) | 38 | 22
Decreased appetite (Metabolism and nutrition disorders) | 112 | 88
Dehydration (Metabolism and nutrition disorders) | 18 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 29 | 29
Hypoalbuminaemia (Metabolism and nutrition disorders) | 23 | 27
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 25 | 23
Hyponatraemia (Metabolism and nutrition disorders) | 35 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 64 | 35
Back pain (Musculoskeletal and connective tissue disorders) | 55 | 36
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 17
Dizziness (Nervous system disorders) | 27 | 21
Headache (Nervous system disorders) | 42 | 33
Neuropathy peripheral (Nervous system disorders) | 12 | 19
Anxiety (Psychiatric disorders) | 19 | 10
Insomnia (Psychiatric disorders) | 24 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 68 | 45
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 67 | 54
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 21 | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 21 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 44 | 36
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 85 | 11
Rash (Skin and subcutaneous tissue disorders) | 76 | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03215706/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT03215706/SAP_001.pdf